CLINICAL TRIAL: NCT01929642
Title: Rapalogues for Autism Phenotype in TSC: A Feasibility Study
Acronym: RAPT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hugo W. Moser Research Institute at Kennedy Krieger, Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AM00037881
Record Dates: First submitted 2013-08-07; First posted 2013-08-28 (Estimated); Results first posted 2021-03-29 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Tuberous Sclerosis Complex; Self-injury; Autism
Keywords: Tuberous Sclerosis Complex (TSC); self-injury; Autism
MeSH Terms: conditions — Tuberous Sclerosis; Self-Injurious Behavior; Autistic Disorder | interventions — Sirolimus; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sirolimus or Everolimus (Experimental): Oral solution or tablet,titrated to therapeutic serum trough range (sirolimus); Oral tablet, titrated to therapeutic serum trough range (everolimus)
  Interventions: Drug: Sirolimus; Drug: Everolimus

INTERVENTIONS:
Drug: Sirolimus
  Other Names: Rapamune, Rapamycin
Drug: Everolimus
  Other Names: Afinitor

SUMMARY:
The purpose of this study is to assess the feasibility and safety of administering rapalogues, sirolimus or everolimus, in participants with Tuberous Sclerosis Complex (TSC) and self-injury and to measure cognitive and behavioral changes, including reduction in autistic symptoms, self-injurious and aggressive behaviors, as well as improvements in cognition across multiple domains of cognitive function.

DETAILED DESCRIPTION:
This is a feasibility and safety study primarily designed to assess the feasibility and safety of conducting a larger clinical trial with sirolimus in individuals with TSC. The present study will employ an ABA design in which three pediatric participants will be selected to receive baseline medical, developmental, behavioral, and cognitive evaluations, followed by a 26 week administration of sirolimus, repeated baseline assessments at the end of the 26 week treatment phase, and a 4 week titrated withdrawal followed by a 22 week period in which no rapalogue is administered. All participants will again be administered baseline medical, behavioral, and cognitive evaluations at the end of the study in order to compare all evaluations done at baseline, the end of the 26 week treatment, and completion of the study. These comparisons will be done to assess secondary outcomes that include reductions in autistic symptoms, self-injury, and aggression, as well as improvements in cognitive function across multiple domains. Furthermore, administration of the secondary outcome measures will also allow us to better understand the sensitivity of these measures in patients with TSC during the course of a clinical trial.

Families of potentially eligible children who express interest in the study and meet prescreening criteria will be invited to attend a screening visit to determine eligibility, inclusion/exclusion criteria, and availability for eight additional study visits. Prior to enrollment, informed consent will be obtained from the parent or legal guardian.

Investigators will use the methods of analysis of single-subject research (ABA design, where first A represents baseline, B represents treatment, and A represents reversal of treatment. The analysis will focus on each of the 3 subjects separately. Data on feasibility and safety (primary outcome) and on frequency of disruptive behavior (secondary outcome) will be plotted and visually inspected to detect any temporal changes by phase: 1. Baseline, 2. Treatment, 3. After treatment. Data in each phase will be summarized as mean +/- standard deviation (SD). We will use the summary data to assess the potential effect of the intervention. Consistency of the effect will be examined across the 3 study participants.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with Tuberous Sclerosis Complex as defined by the revised NIH consensus criteria
2. Possible autism or autism spectrum disorder and/or possible intellectual disability and/or global developmental delay
3. Currently displaying disruptive behaviors, such as self-injury and aggression
4. Seizures or epilepsy with at least one seizure within six months prior to enrollment
5. 2-30 years of age
6. English-speaking caregiver if participant is non-verbal.
7. If individuals are currently being treated with everolimus, they must have been taking it for less than or equal to 6 months.

Exclusion Criteria:

1. Participants who require live vaccines that are contraindicated with sirolimus will be excluded - bacille Calmette Guerin(BCG), measles-mumps-rubella vaccine(MMR), poliovirus, rotavirus, smallpox, typhoid, varicella, or yellow fever.
2. Participants who have a history of multiple or severe infections, or reside in a household with anyone who has a chronic, contagious condition will be excluded. Multiple infections will be defined as eight or more lifetime episodes of otitis media or two or more lifetime episodes of bacterial pneumonia. Severe infections will be defined as infections requiring more than one hospital admission for treatment.
3. Participants with any of the following laboratory abnormalities will be excluded: hematocrit < 27%, absolute neutrophil count(ANC) < 1,500, platelet count < 100,000, serum glutamate oxaloacetate transaminase(SGOT) or serum glutamate pyruvate transaminase (SGPT) > two times normal for age, bilirubin > two times normal for age, alkaline phosphatase > two times normal for age, epidermal growth factor receptor (eGFR) < 30, or evidence of renal failure, hypercholesterolemia.
4. Participants who have medical contraindications to undergoing an MRI will be excluded.
5. Participants with devices implanted in the brain will be excluded.
6. Pregnant participants will be excluded. All young ladies of child bearing potential will have a blood test for pregnancy prior to the start of the study and every study visit for the duration of the study.
7. Participants who have a history of herpes simplex virus, cytomegalovirus, and/or HIV infection will be excluded

Ages: 2 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3 (Actual)
Dates: Start 2013-07; Primary Completion 2016-07 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tanjala Gipson, MD, Principal Investigator — Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Locations (1):
- Kennedy Krieger Institute, Baltimore, Maryland, United States

REFERENCES:
- [Background] Napolioni V, Curatolo P. Genetics and molecular biology of tuberous sclerosis complex. Curr Genomics. 2008 Nov;9(7):475-87. doi: 10.2174/138920208786241243. PMID 19506736
- [Background] Gomez M, Sampson JR, Whittemore VH, editors. Tuberous sclerosis complex. 3rd ed. Oxford University Press; 1999.
- [Background] Osborne JP, Fryer A, Webb D. Epidemiology of tuberous sclerosis. Ann N Y Acad Sci. 1991;615:125-7. doi: 10.1111/j.1749-6632.1991.tb37754.x. No abstract available. PMID 2039137
- [Background] Cross JH. Neurocutaneous syndromes and epilepsy-issues in diagnosis and management. Epilepsia. 2005;46 Suppl 10:17-23. doi: 10.1111/j.1528-1167.2005.00353.x. PMID 16359466
- [Background] Curatolo P, Bombardieri R, Verdecchia M, Seri S. Intractable seizures in tuberous sclerosis complex: from molecular pathogenesis to the rationale for treatment. J Child Neurol. 2005 Apr;20(4):318-25. doi: 10.1177/08830738050200040901. PMID 15921233
- [Background] Joinson C, O'Callaghan FJ, Osborne JP, Martyn C, Harris T, Bolton PF. Learning disability and epilepsy in an epidemiological sample of individuals with tuberous sclerosis complex. Psychol Med. 2003 Feb;33(2):335-44. doi: 10.1017/s0033291702007092. PMID 12622312
- [Background] de Vries PJ. Targeted treatments for cognitive and neurodevelopmental disorders in tuberous sclerosis complex. Neurotherapeutics. 2010 Jul;7(3):275-82. doi: 10.1016/j.nurt.2010.05.001. PMID 20643380
- [Background] Smalley SL. Autism and tuberous sclerosis. J Autism Dev Disord. 1998 Oct;28(5):407-14. doi: 10.1023/a:1026052421693. PMID 9813776
- [Background] Bolton PF, Park RJ, Higgins JN, Griffiths PD, Pickles A. Neuro-epileptic determinants of autism spectrum disorders in tuberous sclerosis complex. Brain. 2002 Jun;125(Pt 6):1247-55. doi: 10.1093/brain/awf124. PMID 12023313
- [Background] Prescibing Information for Sirolimus. 1999).
- [Background] Sindhi R. Sirolimus in pediatric transplant recipients. Transplant Proc. 2003 May;35(3 Suppl):113S-114S. doi: 10.1016/s0041-1345(03)00223-9. PMID 12742479
- [Background] Ehninger D, Han S, Shilyansky C, Zhou Y, Li W, Kwiatkowski DJ, Ramesh V, Silva AJ. Reversal of learning deficits in a Tsc2+/- mouse model of tuberous sclerosis. Nat Med. 2008 Aug;14(8):843-8. doi: 10.1038/nm1788. Epub 2008 Jun 22. PMID 18568033
- [Background] Zeng LH, Xu L, Gutmann DH, Wong M. Rapamycin prevents epilepsy in a mouse model of tuberous sclerosis complex. Ann Neurol. 2008 Apr;63(4):444-53. doi: 10.1002/ana.21331. PMID 18389497
- [Background] Franz DN, Leonard J, Tudor C, Chuck G, Care M, Sethuraman G, Dinopoulos A, Thomas G, Crone KR. Rapamycin causes regression of astrocytomas in tuberous sclerosis complex. Ann Neurol. 2006 Mar;59(3):490-8. doi: 10.1002/ana.20784. PMID 16453317
- [Background] Krueger DA, Care MM, Holland K, Agricola K, Tudor C, Mangeshkar P, Wilson KA, Byars A, Sahmoud T, Franz DN. Everolimus for subependymal giant-cell astrocytomas in tuberous sclerosis. N Engl J Med. 2010 Nov 4;363(19):1801-11. doi: 10.1056/NEJMoa1001671. PMID 21047224
- [Background] Davies DM, de Vries PJ, Johnson SR, McCartney DL, Cox JA, Serra AL, Watson PC, Howe CJ, Doyle T, Pointon K, Cross JJ, Tattersfield AE, Kingswood JC, Sampson JR. Sirolimus therapy for angiomyolipoma in tuberous sclerosis and sporadic lymphangioleiomyomatosis: a phase 2 trial. Clin Cancer Res. 2011 Jun 15;17(12):4071-81. doi: 10.1158/1078-0432.CCR-11-0445. Epub 2011 Apr 27. PMID 21525172
- [Background] Meikle L, Pollizzi K, Egnor A, Kramvis I, Lane H, Sahin M, Kwiatkowski DJ. Response of a neuronal model of tuberous sclerosis to mammalian target of rapamycin (mTOR) inhibitors: effects on mTORC1 and Akt signaling lead to improved survival and function. J Neurosci. 2008 May 21;28(21):5422-32. doi: 10.1523/JNEUROSCI.0955-08.2008. PMID 18495876
- [Background] McCormack FX, Inoue Y, Moss J, Singer LG, Strange C, Nakata K, Barker AF, Chapman JT, Brantly ML, Stocks JM, Brown KK, Lynch JP 3rd, Goldberg HJ, Young LR, Kinder BW, Downey GP, Sullivan EJ, Colby TV, McKay RT, Cohen MM, Korbee L, Taveira-DaSilva AM, Lee HS, Krischer JP, Trapnell BC; National Institutes of Health Rare Lung Diseases Consortium; MILES Trial Group. Efficacy and safety of sirolimus in lymphangioleiomyomatosis. N Engl J Med. 2011 Apr 28;364(17):1595-606. doi: 10.1056/NEJMoa1100391. Epub 2011 Mar 16. PMID 21410393
- [Background] Flaig TW, Costa LJ, Gustafson DL, Breaker K, Schultz MK, Crighton F, Kim FJ, Drabkin H. Safety and efficacy of the combination of erlotinib and sirolimus for the treatment of metastatic renal cell carcinoma after failure of sunitinib or sorafenib. Br J Cancer. 2010 Sep 7;103(6):796-801. doi: 10.1038/sj.bjc.6605868. PMID 20823888
- [Background] Asrani SK, Leise MD, West CP, Murad MH, Pedersen RA, Erwin PJ, Tian J, Wiesner RH, Kim WR. Use of sirolimus in liver transplant recipients with renal insufficiency: a systematic review and meta-analysis. Hepatology. 2010 Oct;52(4):1360-70. doi: 10.1002/hep.23835. PMID 20815021
- [Background] Armstrong AJ, Netto GJ, Rudek MA, Halabi S, Wood DP, Creel PA, Mundy K, Davis SL, Wang T, Albadine R, Schultz L, Partin AW, Jimeno A, Fedor H, Febbo PG, George DJ, Gurganus R, De Marzo AM, Carducci MA. A pharmacodynamic study of rapamycin in men with intermediate- to high-risk localized prostate cancer. Clin Cancer Res. 2010 Jun 1;16(11):3057-66. doi: 10.1158/1078-0432.CCR-10-0124. Epub 2010 May 25. PMID 20501622
- [Background] Habib SL. Tuberous sclerosis complex and DNA repair. Adv Exp Med Biol. 2010;685:84-94. doi: 10.1007/978-1-4419-6448-9_8. PMID 20687497
- [Background] Rapamune: U.S. Physician Prescribing Information. 1999).
- [Background] Krams SM, Martinez OM. Epstein-Barr virus, rapamycin, and host immune responses. Curr Opin Organ Transplant. 2008 Dec;13(6):563-8. doi: 10.1097/MOT.0b013e3283186ba9. PMID 19060543
- [Background] Novak M, Guest C. Application of a multidimensional caregiver burden inventory. Gerontologist. 1989 Dec;29(6):798-803. doi: 10.1093/geront/29.6.798. PMID 2516000
- [Background] Abidin R. Parental stress index - 4, short form. fourth edition ed. Odessa, FL: Psychological Assessment Resources, Inc.; 2009.
- [Background] Staley BA, Montenegro MA, Major P, Muzykewicz DA, Halpern EF, Kopp CM, Newberry P, Thiele EA. Self-injurious behavior and tuberous sclerosis complex: frequency and possible associations in a population of 257 patients. Epilepsy Behav. 2008 Nov;13(4):650-3. doi: 10.1016/j.yebeh.2008.07.010. Epub 2008 Aug 30. PMID 18703161
- [Background] Seizuretracker.com [Internet].; 2012.
- [Background] Roach ES, DiMario FJ, Kandt RS, Northrup H. Tuberous Sclerosis Consensus Conference: recommendations for diagnostic evaluation. National Tuberous Sclerosis Association. J Child Neurol. 1999 Jun;14(6):401-7. doi: 10.1177/088307389901400610. PMID 10385849
- [Background] O'Callaghan FJ, Harris T, Joinson C, Bolton P, Noakes M, Presdee D, Renowden S, Shiell A, Martyn CN, Osborne JP. The relation of infantile spasms, tubers, and intelligence in tuberous sclerosis complex. Arch Dis Child. 2004 Jun;89(6):530-3. doi: 10.1136/adc.2003.026815. PMID 15155396
- [Background] Asano E, Chugani DC, Muzik O, Behen M, Janisse J, Rothermel R, Mangner TJ, Chakraborty PK, Chugani HT. Autism in tuberous sclerosis complex is related to both cortical and subcortical dysfunction. Neurology. 2001 Oct 9;57(7):1269-77. doi: 10.1212/wnl.57.7.1269. PMID 11591847
- [Background] Doherty C, Goh S, Young Poussaint T, Erdag N, Thiele EA. Prognostic significance of tuber count and location in tuberous sclerosis complex. J Child Neurol. 2005 Oct;20(10):837-41. doi: 10.1177/08830738050200101301. PMID 16417883
- [Background] Raznahan A, Higgins NP, Griffiths PD, Humphrey A, Yates JR, Bolton PF. Biological markers of intellectual disability in tuberous sclerosis. Psychol Med. 2007 Sep;37(9):1293-304. doi: 10.1017/S0033291707000177. Epub 2007 Mar 5. PMID 17335641
- [Background] Roid G, Miller L. Leiter international performance scale, revised. Torrance, CA: Western Psychological Services; 1998.
- [Background] Mullen E. Mullen scales of early learning. Circle Pines, MN: American Guidance Service, Inc.; 1995.
- [Background] Wachtel RC, Shapiro BK, Palmer FB, Allen MC, Capute AJ. CAT/CLAMS. A tool for the pediatric evaluation of infants and young children with developmental delay. Clinical Adaptive Test/Clinical Linguistic and Auditory Milestone Scale. Clin Pediatr (Phila). 1994 Jul;33(7):410-5. doi: 10.1177/000992289403300706. PMID 7525138
- [Background] Iwata BA, Pace GM, Kissel RC, Nau PA, Farber JM. The Self-Injury Trauma (SIT) Scale: a method for quantifying surface tissue damage caused by self-injurious behavior. J Appl Behav Anal. 1990 Spring;23(1):99-110. doi: 10.1901/jaba.1990.23-99. PMID 2335488
- [Background] Lord C, Risi S, Lambrecht L, Cook EH Jr, Leventhal BL, DiLavore PC, Pickles A, Rutter M. The autism diagnostic observation schedule-generic: a standard measure of social and communication deficits associated with the spectrum of autism. J Autism Dev Disord. 2000 Jun;30(3):205-23. PMID 11055457
- [Background] Lord C, Rutter M, Le Couteur A. Autism Diagnostic Interview-Revised: a revised version of a diagnostic interview for caregivers of individuals with possible pervasive developmental disorders. J Autism Dev Disord. 1994 Oct;24(5):659-85. doi: 10.1007/BF02172145. PMID 7814313
- [Background] Constantino J. The social responsiveness scale. Los Angeles: Western Psychological Services; 2002.
- [Background] Rutter M, Bailey A, Lord C. Social communication questionnaire. Western Psychological Services; 2003.
- [Background] Granader YE, Bender HA, Zemon V, Rathi S, Nass R, Macallister WS. The clinical utility of the Social Responsiveness Scale and Social Communication Questionnaire in tuberous sclerosis complex. Epilepsy Behav. 2010 Jul;18(3):262-6. doi: 10.1016/j.yebeh.2010.04.010. PMID 20554253
- [Background] Mirenda P, Smith IM, Vaillancourt T, Georgiades S, Duku E, Szatmari P, Bryson S, Fombonne E, Roberts W, Volden J, Waddell C, Zwaigenbaum L; Pathways in ASD Study Team. Validating the Repetitive Behavior Scale-revised in young children with autism spectrum disorder. J Autism Dev Disord. 2010 Dec;40(12):1521-30. doi: 10.1007/s10803-010-1012-0. PMID 20405194
- [Background] Kazdin AE. Single-case research designs in clinical child psychiatry. J Am Acad Child Psychiatry. 1983 Sep;22(5):423-32. doi: 10.1016/s0002-7138(09)61503-x. No abstract available. PMID 6630801
- [Background] Sanchez CP, He YZ. Bone growth during rapamycin therapy in young rats. BMC Pediatr. 2009 Jan 13;9:3. doi: 10.1186/1471-2431-9-3. PMID 19144108
- [Background] Alvarez-Garcia O, Carbajo-Perez E, Garcia E, Gil H, Molinos I, Rodriguez J, Ordonez FA, Santos F. Rapamycin retards growth and causes marked alterations in the growth plate of young rats. Pediatr Nephrol. 2007 Jul;22(7):954-61. doi: 10.1007/s00467-007-0456-8. Epub 2007 Mar 17. PMID 17370095
- [Background] Rangel GA, Ariceta G. Growth failure associated with sirolimus: case report. Pediatr Nephrol. 2009 Oct;24(10):2047-50. doi: 10.1007/s00467-009-1215-9. Epub 2009 Jun 3. PMID 19495804
- See also: Kennedy Krieger Institute Clinical Trials Unit — http://www.kennedykrieger.org/research-training/participate-in-research/clinical-trials
- See also: TSC clinic at Kennedy Krieger Institute — http://www.kennedykrieger.org/patient-care/patient-care-programs/outpatient-programs/tuberous-sclerosis-clinic

RESULTS

PARTICIPANT FLOW:
Groups:
- Sirolimus or Everolimus: Oral solution or tablet,titrated to therapeutic serum trough range (sirolimus); Oral tablet, titrated to therapeutic serum trough range (everolimus)
  Sirolimus
  Everolimus
Period: Overall Study
Arm/Group | Sirolimus or Everolimus
Started | 3
Completed | 1
Not Completed | 2

BASELINE CHARACTERISTICS:
Groups:
- Everolimus or Sirolimus: Medication choice
Arm/Group | Everolimus or Sirolimus
Number analyzed (Participants) | 3
Age, Continuous [Mean (Full Range); unit: years] | 7 [3 to 13]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Compliance to the Treatment Protocol.
Description: One outcome measurement of feasibility will include family/patient compliance with the treatment protocol, which will be assessed and documented at every study visit and telephone follow-up call, by the physician and/or study team member. This was calculated by calculating dividing the total number of study visits and study assessments completed by the total number of study visits and study assessments indicated by the treatment protocol.
Time Frame: Change from baseline to EOT visit 12 week 53
Measure: Number; unit: percentage of completed visits/measures
Groups:
- Everolimus or Sirolimus: Medication
Arm/Group | Everolimus or Sirolimus
Number analyzed (Participants) | 3
percentage of completed visits/measures
  Participant 002 | 100
  Participant 003 | 58
  Participant 001 | 58

2. Primary Outcome: Caregiver Burden
Description: The Caregiver Burden Scale is a standard set of questions which will be used to measure the non-medical impact of TSC on caregivers and how it affects the feasibility of study completion.
  The Caregiver's Burden Scale (CBS) is a 22-item scale that assess subjectively experienced burden by caregiver's to chronically disabled persons. maximum scores: 88 & Minumum scores: 22
  High values represent a worse outcome
Time Frame: Change from baseline to EOT visit 12 week 53
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Everolimus or Sirolimus
Number analyzed (Participants) | 3
units on a scale | 61 [45 to 70]

3. Primary Outcome: Feasibility Measurements of Parental Stress
Description: Measurements of stress will be administered. Specifically, we will use the Parental Stress Index. Quantifying stress, as well as compliance with the study protocol, will allow investigators to objectively assess the feasibility of a larger clinical trial of sirolimus in patients with TSC.
  Parental stress index maximum score: 180 Parental stress index minimum score: 36 higher raw scores indicate higher levels of stress.
Time Frame: Change from baseline to EOT visit 12 week 53
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Everolimus or Sirolimus
Number analyzed (Participants) | 3
units on a scale | 111 [86 to 132]

4. Secondary Outcome: Total Number of Aggressions or Self-injuries
Description: This is the total number of aggressions or self-injuries for all participants.
Time Frame: 1 year
Measure: Number; unit: Number of aggressions or self-injuries
Arm/Group | Everolimus or Sirolimus
Number analyzed (Participants) | 3
Number of aggressions or self-injuries | 82

5. Secondary Outcome: Cognitive Function as Assessed by the Capute Scale
Description: Score range maximum: 100 Score range minimum: 0
  High values represent a high cognitive function Below 70 is abnormal. 70-100 is the normal range.
Time Frame: 1 year
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Everolimus or Sirolimus
Number analyzed (Participants) | 3
score on a scale | 15 [14 to 21]

6. Secondary Outcome: Repetitive Behavior
Description: Repetitive behavior will be assessed using the Repetitive Behavior Scale - revised, a questionnaire to characterize several domains of repetitive behavior including ritualistic behavior, stereotypic behavior, self-injurious behavior, compulsive behavior, and restricted interests.
  There are 36 items on the scale. Behaviors are rated on a 4-point scale: 0-Behavior does not occur, 1-Behavior occurs and is a mild problem, 2-Behavior occurs and is a moderate problem, 3-Behavior occurs and is a severe problem.
  Maximum score: 108 & minimum score: 0 A high score represents the worse outcome
Time Frame: 1 year
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Everolimus or Sirolimus
Number analyzed (Participants) | 3
score on a scale | 69 [58 to 80]

7. Secondary Outcome: Self-Injury Trauma Scale--SIT Scale
Description: The SIT Scale is a 3-part clinician-completed scale used to quantify visible injuries caused by self-injurious behavior(SIB). Part 1 includes sections to indicate SIB topographies and any evidence of healed injury. In Part 2 evaluators document the location and severity of injury (on a 3-point scale). In Part 3, respective scores from Parts 1 and 2 are summed to obtain a Number Index, a Severity Index, and Estimate of Current Risk. This Scale has been used in research with adults with SIB with inter-rater reliability averaging 85%.
  Maximum score: 100 Minimum score: 0 High score represent worse outcome.
Time Frame: 1 year
Population: Self-injury was not severe enough to use the scale. Therefore analysis was not done.
Arm/Group | Everolimus or Sirolimus
Number analyzed (Participants) | 0

8. Secondary Outcome: Frequency of Seizures Assessed by Total Number of Seizures
Description: Parents will be asked to document the frequency of their child's seizures using a manual or electronic (seizuretracker.com) seizure diary. The total number of seizures at baseline for all participants.
Time Frame: at baseline
Measure: Number; unit: seizures
Arm/Group | Everolimus or Sirolimus
Number analyzed (Participants) | 3
seizures | 0

ADVERSE EVENTS:
Arm/Group | Everolimus
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 1/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Everolimus (N=3)
aphthous ulcer (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No